CLINICAL TRIAL: NCT04784793
Title: A Mobile App for Postural Alignment Exercises in Cervical and Thoracic Spine Regions: Design, Development, Usability and Randomized Controlled Pilot Study
Brief Title: Postural Alignment Exercise Mobile App for Cervical and Thoracic Spine Regions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Marmara University, Scientific Research Projects Committee (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09.2018.069
Record Dates: First submitted 2021-02-28; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Development and Design of Mobile App; Preventive Physiotherapy; Exercise Adherence; Cervical and Thoracic Spine
Keywords: mHealth; Postural alignment; Preventive physiotherapy; Exercise adherence; Neck pain; Upper back pain
MeSH Terms: conditions — Neck Pain; Back Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase1: Design and development (No Intervention): We conducted focus group meetings to discuss the content, features and design of the app.
  The focus group consisted of physiotherapists and young adults. The focus group members discussed the variety of topics in subgroups (login parameters, self-monitoring, exercises content, video or animation types, exercise diary, reminders, encouragement, method, etc).
- Phase 2: Testing the app (No Intervention): We tested the prototype version app interface in the 2nd phase. All participants downloaded the prototype app and used the app for one week.
- Phase 3: Usability evaluation (No Intervention): We conduct a think-aloud interview and evaluate the quantitative usability in the third phase.
  The quantitative usability was assessed by the System Usability Scale (SUS), and the adapted Usability, Satisfaction and Ease to Use (USE) Questionnaire.
- Phase 4: Pilot randomized controlled trial/ The app-based group (Active Comparator): The app-based group:
  Participants in the intervention group received their smartphone-based- home exercise program.
  Interventions: Other: App-based group
- Phase 4: Pilot randomized controlled trial/ The control group (Experimental): The control group:
  Participants in the control group received their home exercise programs as a paper handout.
  Interventions: Other: Control group

INTERVENTIONS:
Other: App-based group — Participants received home exercise programs by a postural alignment exercise mobile app we developed.
  The postural alignment app included 3 main emerged themes were recorded as self-assessment, neck/shoulder, and upper back-specific exercise content, and motivational notifications.
  Participants can evaluate themselves in the application thanks to the self-assessment, receive motivational notifications during the day, and exercise reminders on the days determined by them. They can apply the exercise program with the formed exercise content videos.
  The exercise program consists of combined exercises that postural alignment plus exercises of neck spinal stabilization, stretching, and strengthening of neck/shoulders/upper back regions.
  Both group participants were requested to do the exercises from the app/brochure 3 times a week, for 6 weeks.
  Arms: Phase 4: Pilot randomized controlled trial/ The app-based group
Other: Control group — Participants received home exercise programs as a paper handout.
  The exercise program was the same for app-based and control groups.
  Both group participants were requested to do the exercises from the app/brochure 3 times a week, for 6 weeks.
  Arms: Phase 4: Pilot randomized controlled trial/ The control group

SUMMARY:
Postural alignment in the cervical and thoracic regions is affected by various risks such as smartphone use in particular young adults. The small screen of smartphones causes ergonomic risk for posture and musculoskeletal system. Previous studies found that neck, shoulder, and upper back pain associated with the overuse of smartphones. Neck pain often arises from unideal postures. Participants should be informed about these risks and encouraged to exercise to be protective. Digital health apps' use is rising by the day and health apps offer opportunities for both healthcare professionals and users.

Therefore, this study aimed to develop an app including preventive exercise interventions to keep postural alignment in cervical and thoracic spine regions employing an iterative, user-centred design and to test the usability of the app and evaluate its effectiveness with a pilot randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* to be a university student aged 18-25, to be a smartphone user for more than 3 years with more than three hours daily use.

Exclusion Criteria:

* if they had any chronic health problems (rheumatic, orthopedic, neurological, cardiopulmonary, vestibular system), any trauma in the neck/upper back/upper limb region in the last six months, had a congenital deformity, had received another treatment or having surgery in last one year.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of musculoskeletal problems | Baseline
  Musculoskeletal problems were assessed by Nordic Musculoskeletal Questionnaire. The Nordic Musculoskeletal Questionnaire queries yes/no for nine body regions so far, in the last 12 months, and in the last 7 days of evaluation, whether ache, pain, or discomfort.
VAS | Baseline and at end of the 6 weeks
  Neck pain was assessed by Visual Analog Scale (VAS) before and after the 6 weeks exercise program. The participants were instructed to mark a point on a line between zero (no pain) and 10 cm (maximum pain).
Neck Pain and Disability Scale | Baseline and at end of the 6 weeks
  Functional disability associated with neck pain was evaluated by the Neck Pain and Disability Scale (NPAD) questionnaire before and after the 6 weeks exercise program. The Neck Pain and Disability Scale consists of 20 items and each item was scored from 0 to 5, and the total score is the sum of the item scores [possible range 0 (no pain)-100 (maximal pain)].

SECONDARY OUTCOMES:
Evaluation of exercise adherence | At end of the 6 weeks
  The app automatically gathers total usage status (count of participated sessions, usage times) when participants login to the app to start an exercise program.
  Exercise adherence was measured with a ratio of total participated sessions compared with the target defined.
Evaluation of app satisfaction | At end of the 6 weeks
  Users were evaluated to rate their satisfaction with the intervention on a 5-point Likert scale after 6 weeks period.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Tonga, PHD, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim HJ; DH; Kim JS. The relationship between smartphone use and subjective musculoskeletal symptoms and university students. J Phys Ther Sci. 2015 Mar;27(3):575-9. doi: 10.1589/jpts.27.575. Epub 2015 Mar 31. PMID 25931684
- [Result] Slater H, Stinson JN, Jordan JE, Chua J, Low B, Lalloo C, Pham Q, Cafazzo JA, Briggs AM. Evaluation of Digital Technologies Tailored to Support Young People's Self-Management of Musculoskeletal Pain: Mixed Methods Study. J Med Internet Res. 2020 Jun 5;22(6):e18315. doi: 10.2196/18315. PMID 32442143
- [Result] Stutz T, Emsenhuber G, Huber D, Domhardt M, Tiefengrabner M, Oostingh GJ, Fotschl U, Matis N, Ginzinger S. Mobile Phone-Supported Physiotherapy for Frozen Shoulder: Feasibility Assessment Based on a Usability Study. JMIR Rehabil Assist Technol. 2017 Jul 20;4(2):e6. doi: 10.2196/rehab.7085. PMID 28729234
- [Result] Toelle TR, Utpadel-Fischler DA, Haas KK, Priebe JA. App-based multidisciplinary back pain treatment versus combined physiotherapy plus online education: a randomized controlled trial. NPJ Digit Med. 2019 May 3;2:34. doi: 10.1038/s41746-019-0109-x. eCollection 2019. PMID 31304380
- [Result] Xie Y, Szeto G, Dai J. Prevalence and risk factors associated with musculoskeletal complaints among users of mobile handheld devices: A systematic review. Appl Ergon. 2017 Mar;59(Pt A):132-142. doi: 10.1016/j.apergo.2016.08.020. Epub 2016 Sep 11. PMID 27890121